CLINICAL TRIAL: NCT03265574
Title: Preventing Cardiac Damage in Patients Treated for Breast Cancer and Lymphoma: a Phase 3 Randomised, Open Label, Blinded Endpoint, Superiority Trial of Enalapril to Prevent Anthracycline-induced CardioToxicity
Brief Title: PROACT: Can we Prevent Chemotherapy-related Heart Damage in Patients With Breast Cancer and Lymphoma?
Acronym: PROACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: South Tees Hospitals NHS Foundation Trust (Other)
Collaborators: Newcastle University (Other); University of Durham (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016152
Record Dates: First submitted 2017-08-24; First posted 2017-08-29 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Non Hodgkin Lymphoma
MeSH Terms: conditions — Breast Neoplasms; Lymphoma, Non-Hodgkin | interventions — Enalapril

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Drug: Enalapril
- Standard care (No Intervention)

INTERVENTIONS:
Drug: Enalapril — Enalapril is an Angiotensin Converting Enzyme (ACE) inhibitor which supresses the reninangiotensin-aldosterone system resulting in increased plasma renin activity and decreased aldosterone secretion
  Arms: Intervention

SUMMARY:
PROACT will establish the effectiveness of the angiotensin-converting enzyme inhibitor (ACEI) enalapril maleate (enalapril) in preventing cardiotoxicity in patients with breast cancer and non-Hodgkin lymphoma undergoing adjuvant epirubicin-based chemotherapy.

DETAILED DESCRIPTION:
PROACT is a phase 3 randomised, open label, blinded endpoint, superiority trial of enalapril to prevent anthracycline-induced in patients treated for breast cancer and lymphoma.

Anthracyclines used in the treatment of breast cancer cause damage to heart muscle cells; this results in cell death (cardiotoxicity). In UK contemporary practice, epirubicin is the most frequently used anthracycline.

Patients due to receive adjuvant anthracycline chemotherapy (planned epirubicin dose >300mg/m2) for breast cancer at four specialist centres in the North of England will be invited to participate. 170 eligible patients will be randomised in a 1:1 ratio, to either enalapril plus usual care or to usual care. Enalapril will be commenced prior to the first anthracycline dose, titrated to a maximum tolerated dose, and continued during chemotherapy. Chemotherapy will continue per usual care; typically six treatment cycles. Patients will have a blood test performed at the end of each chemotherapy cycle to measure cardiac troponin, and at one month following the last epirubicin dose. Investigators and patients will be blinded to the troponin results. Patients will have an echocardiogram at baseline and following their chemotherapy; they will be assessed in a blinded manner by a central Core Laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Adult patients with histopathologically* confirmed breast carcinoma who have received surgery for their breast cancer; planned to receive 6 cycles of EC 90 (total planned dose 540mg/m2 epirubicin) or FEC 75 (total planned dose 450mg/m2 epirubicin) adjuvant chemotherapy regimen. Patients with HER2+ breast cancer are eligible for inclusion.

OR

* Adult patients with histopathologically confirmed non-Hodgkin lymphoma (NHL), planned to receive 6 cycles of R-CHOP or CHOP (total planned dose 300mg/m2 doxorubicin) chemotherapy**

  * Patients with HER2+ breast cancer are eligible for inclusion. ** Patients who will receive an alternative anti-CD20 monoclonal antibody are eligible (for example O-CHOP), as long as the total planned doxorubicin dose is ≥300mg/m2 over 6 cycles

Exclusion Criteria:

* Positive baseline cardiac troponin T (≥14ng/L);
* known contraindication to ACE inhibitor e.g. renal artery stenosis, severe aortic stenosis;
* are taking, or have a previous intolerance to ACEI (e.g. angioedema);
* patient already taking other agents acting on the renin-angiotensin-aldosterone system e.g. Aliskiren, angiotensin receptor blockers (ARBs), Entresto (sacubitril/valsartan), spironolactone, eplerenone;
* LVEF <50%*;
* estimated GFR < 30 mL/min/1.73m2 at baseline;
* hyperkalaemia defined as serum potassium ≥5.5mmol/L;
* symptomatic hypotension, or Systolic Blood Pressure <100mmHg;
* poorly-controlled hypertension (Blood Pressure >160/100mmHg**, or ambulatory BP of 150/95mmHg);
* previous myocardial infarction;
* known metastatic breast cancer;
* previous exposure to anthracycline chemotherapy;
* are pregnant or breastfeeding;
* previous Herceptin treatment or planned Herceptin treatment within four weeks following anthracycline chemotherapy;
* for patients of childbearing potential: refusal to use adequate contraception throughout the trial;***
* any other invasive cancer diagnosed and treated in the past 5 years;
* symptomatic or severe asymptomatic radiation-induced cardiac disease;
* judgement by the investigator that the patient has a prognosis of < 1 year or are unlikely to complete 6 cycles of chemotherapy;
* judgement by the investigator that the patient is high risk for tumour lysis syndrome (applicable only to NHL patients);
* judgement by the Investigator that the patient should not participate in the study, for example, if the patient is unlikely to comply with study procedures, restrictions, and requirements.

  *<50% as defined by Simpson's biplane method; if absolute measurements are not possible, then a visually normal assessment of LVEF is acceptable for inclusion.

  **White coat hypertension is more common, and should be ruled out by an ambulatory blood pressure monitor

  ***Female patients between the ages of 18 and 50 will receive a pregnancy test at baseline. Adequate methods of contraception are those that can achieve a failure rate of less than

  1% per year when used consistently and correctly, such methods include:
* combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation

  * oral
  * intravaginal
  * transdermal
* progestogen-only hormonal contraception associated with inhibition of ovulation

  * oral
  * injectable
  * implantable
* intrauterine device (IUD)
* intrauterine hormone-releasing system (IUS)
* bilateral tubal occlusion
* vasectomy/vasectomised partner
* true sexual abstinence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Cardiac troponin T release | One month after last dose of anthracycline
  Cardiac troponin T release during anthracycline treatment

SECONDARY OUTCOMES:
Cardiac function | One month after last dose of anthracycline
  Cardiac function assessed by echocardiogram
Adherence to enalapril | One month after last dose of anthracycline
  Ability of participant to adhere to enalapril
Adverse Events / Reactions | One month after last dose of anthracycline
  Number and severity of Adverse Events and Reactions
Anxiety or distress related to trial participation | One month after last dose of anthracycline
  Anxiety or distress related to trial participation
Cancer and chemotherapy outcomes | One month after last dose of anthracycline
  Cancer and chemotherapy outcomes in the population under study
Cardiac troponin I release | One month after last dose of anthracycline
  cardiac troponin I release during anthracyline treatment

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Hildreth, Study Chair — Study Chair
Locations (1):
- South Tees Hospitals NHS FT, Middlesbrough, Teesside, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Austin D, Maier RH, Akhter N, Sayari M, Ogundimu E, Maddox JM, Vahabi S, Humphreys AC, Graham J, Oxenham H, Haney S, Cresti N, Verrill M, Osborne W, Wright KL, Goranova R, Bailey JR, Kalakonda N, Macheta M, Kilner MF, Young ME, Morley NJ, Neelakantan P, Gilbert G, Thomas BK, Graham RJ, Fujisawa T, Mills NL, Hildreth V, Prichard J, Kasim AS, Hancock HC, Plummer C. Preventing Cardiac Damage in Patients Treated for Breast Cancer and Lymphoma: The PROACT Clinical Trial. JACC CardioOncol. 2024 Aug 27;6(5):684-696. doi: 10.1016/j.jaccao.2024.07.010. eCollection 2024 Oct. PMID 39479329
- [Derived] Maier RH, Plummer C, Kasim AS, Akhter N, Ogundimu E, Maddox J, Graham J, Stewart M, Wardley A, Haney S, Vahabi S, Oxenham H, Humphreys A, Cresti N, Verrill M, Graham R, Chang L, Hancock HC, Austin D. Preventing cardiotoxicity in patients with breast cancer and lymphoma: protocol for a multicentre randomised controlled trial (PROACT). BMJ Open. 2022 Dec 30;12(12):e066252. doi: 10.1136/bmjopen-2022-066252. PMID 36585130